CLINICAL TRIAL: NCT03584438
Title: The Effects of Theta-Burst Stimulation Duration on Human Motor Cortex Excitability
Brief Title: iTBS Methods and Motor Cortex Excitability
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: MUSC Center for Biomedical Research Excellence in Stroke Recovery (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 68775
Record Dates: First submitted 2018-06-15; First posted 2018-07-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Motor Activity
Keywords: TMS; Motor Cortex; Excitability; LTP; LTD
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 30 healthy controls will undergo four Active TMS treatment sessions (separated by at least 24 hrs), along with a Sham TMS treatment session. The theta-burst treatments will be counterbalanced across participants.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Hanlon Real iTBS Protocol 1 (Experimental): One session of real intermittent Theta Burst Stimulation (iTBS) will be delivered to the left motor cortex. 600 pulses of iTBS over the motor cortex (C3), 3600 pulses are delivered over 19 minutes.
  Interventions: Device: Real iTBS
- Hanlon Real iTBS Protocol 2 (Experimental): One session of real intermittent Theta Burst Stimulation (iTBS) will be delivered to the left motor cortex. 600 pulses of iTBS over the motor cortex (C3), 1800 pulses are delivered over 9 minutes and 30 seconds.
  Interventions: Device: Real iTBS
- Huang Real iTBS Protocol (Experimental): One session of real intermittent Theta Burst Stimulation (iTBS) will be delivered to the left motor cortex. (2 sec trains of tbs every 10 sec) was applied over the left motor cortex (C3) for 190 seconds (a total of 600 TMS pulses).
  Interventions: Device: Real iTBS
- Gamboa Real iTBS Protocol (Experimental): One session of real intermittent Theta Burst Stimulation (iTBS) will be delivered to the left motor cortex. (2 sec trains of tbs every 10 sec) was applied over the left motor cortex (C3) for 380 seconds (a total of 1200 TMS pulses).
  Interventions: Device: Real iTBS
- Sham iTBS protocol (Sham Comparator): One session of sham intermittent Theta Burst Stimulation (iTBS) will be delivered to the left motor cortex. The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin over the left motor cortex (C3) and beneath the coil.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Real iTBS — This will be delivered with the Magventure Magpro system; pulses are delivered with the active coil (double blinded using the Universal Serial Bus key)
  Arms: Gamboa Real iTBS Protocol; Hanlon Real iTBS Protocol 1; Hanlon Real iTBS Protocol 2; Huang Real iTBS Protocol
Device: Sham iTBS — This will be delivered with the Magventure Magpro system; pulses are delivered with the sham coil (double blinded using the Universal Serial Bus key). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham iTBS protocol

SUMMARY:
In a recent publication by Gamboa et al. 20108 it was shown that extended theta-burst stimulation duration might have reverse effects on cortical excitability when compared to the original Huang et al. 2005 publication. While the post treatment effects of the original Huang et al. 2005 protocol were successfully replicated, when continuous theta burst stimulation (cTBS) protocols were doubled to 1200 pulses over 80 seconds and the iTBS protocols were doubled to 1200 pulses over 390 seconds, there was increased facilitation after the prolonged cTBS and decreased excitability after prolonged iTBS. Currently there is an interest in optimizing repetitive transcranial magnetic stimulation (rTMS) protocols and in particular theta burst stimulation as both a therapeutic and an investigational tool. In Hanlon et al. 2015, a novel theta burst paradigm is described in which two trains of 1800 pulses of cTBS were administered, each train separated by a one-minute interval. In this study 11-cocaine dependent individuals underwent cTBS over the medial prefrontal cortex (MPFC) and showed attenuated craving as well as decreases in activity of the striatum and anterior insula. This study aims to replicate the findings of the Gamboa and Huang protocols as well as investigate how novel theta burst stimulation paradigms such as those described in Hanlon et al. 2015, which are currently being explored as therapeutic methods in addiction may change cortical excitability.

DETAILED DESCRIPTION:
rTMS is a method of non-invasive neuromodulation. Although TMS (transcranial magnetic stimulation) has widely been used as a research method to better understand brain neurophysiology, rTMS protocols have been shown to be clinically beneficial to patients suffering from neurological disorders such as Parkinson's Disease and stroke as well as psychiatric diseases such as major depression. In October of 2008 the FDA approved 10 Hertz (Hz) dorsolateral prefrontal cortex (DLPFC) stimulation for patients with medication resistant depression. The typical duration of a single rTMS treatment for depression lasts for about 30 minutes, but must be repeated daily over several weeks. The decision to use DLPFC stimulation was due in part to imaging studies, which suggested depressed patients had decreased activity in the region. Thus, rTMS could be used to reverse those behavioral effects of depression by increasing activity in the DLPFC. Traditionally 5 Hertz (Hz) stimulation and upward has been shown to be excitatory while stimulation of 0.2-1 Hertz (Hz) has been shown to have inhibitory effects on the cortex. Although these parameters appear to be efficacious the development of new rTMS methods are still being explored.

Theta burst stimulation (TBS) is a method with the potential of providing excitatory or inhibitory effects on the cortex, which are as powerful as traditional rTMS methods yet more efficient in duration and intensity required. Evidence from previous studies looking at theta burst as a treatment for depression has highlighted the importance of the method's development. One study indicated that theta-burst stimulation over the dorsomedial prefrontal cortex (DMPFC) for a duration of just 6 minutes can produce comparable anti-depressant effects to traditional 10Hz stimulation over 30 minutes. Theta burst stimulation effects were first empirically tested on the human motor cortex by Huang et al. 2005. The effects of stimulation (80% of active motor threshold) over the motor cortex were measured pre and post treatment with electromyography (EMG) recordings of motor evoked potentials (MEPs) on a small contralateral hand muscle in response to single pulses of TMS. Two protocols showed changes in excitability of the corticospinal tract, including cTBS defined as three burst stimuli at 50 Hz with 20ms between stimuli repeated every 200ms at 5Hz and iTBS defined as a 2s train of TBS repeated every 10 seconds. Although both protocols deliver a total of 600 pulses, the cTBS protocols lasts for 40 seconds while the iTBS protocol lasts for 190 seconds. Huang et al. 2005 determined that cTBS over motor cortex decreased excitability while iTBS increased excitability which were present an hour following treatment.

The excitability of the motor cortex may be modulated differently depending on the type of theta burst stimulation protocol utilized. iTBS was originally described by Huang et al. 2005 resulting in an excitatory effects (LTP like) on the cortex. Gamboa et al. 2010 later confirmed this finding but showed that there was a decrease in excitability (LTD-like) when the protocol is doubled. Both of these protocols are to be replicated and in addition 2 new protocols. In order to investigate how cortical excitability changes as a function of protocol, MEPs will be recorded using EMG on the hand muscle contralateral to the stimulated cortex. Baseline MEPs will be obtained pretreatment, followed by one of the four theta burst protocols, or a sham treatment. Theta burst protocols are to be administered to each participant in randomized order. After theta burst is administered 20 MEPs will be collected at 0, 10, 20, 30, 40, 50 and 60 minutes.

Specific Aim 1: To determine the long-term potentiation (LTP) like and long-term depression (LTD) like effects of four different theta burst stimulation protocols on motor cortex excitability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (18 - 65 years of age)
* Able to read and understand questionnaires and informed consent

Exclusion Criteria:

* Pregnancy, females of child bearing age must undergo a pregnancy test to confirm eligibility;
* History of seizure disorder or post-stroke seizure;
* Implanted medical devices or metal in head (except braces);
* Preexisting scalp lesion or wound or bone defect or hemicraniectomy;
* Left-hand dominance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-26 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Effects of theta burst stimulation protocols of LTP-like and LTD-like stimulation on change in motor cortex excitability | Through study completion, an average of two weeks.
  The excitability of the motor cortex may be modulated differently depending on the type of TBS protocol utilized. iTBS was originally described by Huang et al. 20057 resulting in an excitatory effects (LTP like) on the cortex. Gamboa et al. 20108 later confirmed this finding but showed that there was a decrease in excitability (LTD-like) when the protocol is doubled. Both of these protocols are to be replicated and in addition 2 new protocols. In order to investigate how cortical excitability changes as a function of protocol, MEPs (motor evoked potentials) will be recorded using EMG (electromyography) on the hand muscle contralateral to the stimulated cortex. Baseline MEPs will be obtained pretreatment, followed by one of the four theta burst protocols, or a sham treatment. Theta burst protocols are to be administered to each participant in randomized order. After theta burst is administered 20 MEPs will be collected at 0, 10, 20, 30, 40, 50 and 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McTeague, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No